CLINICAL TRIAL: NCT07267897
Title: The Effect of Preoperative Nebulized Lidocaine and Nebulized 3% NaCl Premedication on Postoperative Respiratory Complications in Pediatric Patients Undergoing Adenoidectomy and/or Adenotonsillectomy Surgery
Brief Title: Nebulized Lidocaine vs 3% Sodium Chloride in Pediatric Adenoid/Tonsil Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Burçin Alaçam, MD, medicine doctor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SAU-ANE-BA-01
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Respiratory Complication
Keywords: Postoperative Respiratory Complication; Lidocaine; %3 Sodium Chloride; Pediatric; Adenoidectomy; Adenotonsillectomy
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design in which pediatric patients undergoing adenoidectomy and/or adenotonsillectomy are randomly assigned to one of the intervention groups. Each participant will receive only one type of preoperative nebulized treatment (lidocaine, 3% hypertonic saline, or control), and outcomes will be compared between the groups throughout the study period.
Who Masked: Participant, Care Provider
Masking Description: This study is double-blinded. Both the participants and the care providers administering the nebulized treatment will be unaware of the group assignments. The nebulized solutions (lidocaine, 3% hypertonic saline, or control) will be prepared in identical containers with identical appearance to ensure blinding throughout the perioperative period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup L (Experimental): Patients will receive 0.2 ml/kg of nebulized lidocaine under monitoring, with the treatment completed 15 minutes prior to the surgical procedure.
  Interventions: Drug: Nebulize Lidocaine
- Grup H (Experimental): Patients will receive 0.2 ml/kg of nebulized %3 hypertonic saline under monitoring, with the treatment completed 15 minutes prior to the surgical procedure..
  Interventions: Drug: Nebulize %3 Sodium Chloride

INTERVENTIONS:
Drug: Nebulize Lidocaine — Preoperative administration of lidocaine via nebulization at 0.2 ml/kg to reduce postoperative respiratory complications.
  Other Names: Lidocaine
  Arms: Grup L
Drug: Nebulize %3 Sodium Chloride — Preoperative administration of 3% hypertonic saline via nebulization at 0.2 ml/kg to reduce postoperative respiratory complications.
  Other Names: %3 NaCl
  Arms: Grup H

SUMMARY:
This prospective, randomized clinical trial aims to evaluate the effect of preoperative nebulized lidocaine and nebulized 3% hypertonic sodium chloride (NaCl) on the incidence of postoperative respiratory complications in pediatric patients undergoing adenoidectomy and/or adenotonsillectomy. Lidocaine, a versatile sodium channel blocker, has shown antitussive, bronchodilatory, and anti-inflammatory benefits when nebulized, and has been safely used in children for respiratory procedures. Hypertonic 3% NaCl is known to improve mucociliary clearance, reduce airway edema, and enhance secretion mobilization, particularly in pediatric respiratory conditions. Both agents have demonstrated individual safety and efficacy in respiratory management, yet their preoperative nebulized use for preventing postoperative respiratory adverse events (PRAEs) in pediatric airway surgery has not been previously studied. This trial seeks to determine whether preoperative nebulization with these agents can reduce postoperative respiratory complications, improve recovery, and enhance perioperative safety in this high-risk population.

DETAILED DESCRIPTION:
Lidocaine is a drug with multiple clinical uses. Beyond its classical indication as a sodium channel blocker in local, regional, and neuraxial anesthesia, it has been:

* administered intravenously as an antitussive agent in ophthalmic surgery,
* used in both human and veterinary anesthesia to reduce the minimum alveolar concentration (MAC),
* applied as an analgesic for acute pain,
* used as an antiarrhythmic for ventricular arrhythmias,
* administered as a cardioplegic agent in cardiac surgery,
* used as a local anesthetic for venous cannulation,
* nebulized during awake airway interventions,
* nebulized in refractory cough, and
* applied into the endotracheal tube cuff to prevent postoperative sore throat.

Nebulized lidocaine has previously been used in adults with chronic obstructive pulmonary disease, acute asthma, and acute lung infections to suppress cough and provide bronchodilation, and has been found safe and effective. High doses (up to 8 mg/kg) of nebulized lidocaine have been safely administered in infants and children prior to flexible bronchoscopy to reduce perioperative respiratory adverse events (PRAEs).

Hypertonic 3% sodium chloride (NaCl) solution is an agent that has been extensively studied and used clinically in respiratory diseases. Its primary mechanisms of action include osmotic rehydration of the airway surface liquid, thinning mucus, and facilitating mucociliary clearance. This reduces secretion viscosity and supports easier mucus removal. It may also reduce airway edema, relieve obstruction, and promote the dissolution of mucus plugs. Some studies suggest it may exert anti-inflammatory effects by limiting inflammatory mediators. In clinical practice, it has been shown to be safe and effective in children with acute bronchiolitis, reducing hospital stay and improving symptoms. In addition, it is used in cystic fibrosis, chronic bronchitis, COPD, and acute pulmonary infections to enhance mucus clearance and improve respiratory function.

Adenoidectomy and tonsillectomy are among the most common surgical procedures performed in the pediatric population, primarily due to recurrent throat infections and sleep-disordered breathing associated with obstructive sleep apnea. Postoperative complications may include bleeding, respiratory distress, airway obstruction, postoperative pain, and dehydration. Reported respiratory complication rates range from 2% to 4%, rising to 13-15% in high-risk groups. Beyond the inherent respiratory risks of the surgery itself, perioperative respiratory adverse events (PRAEs) are highly prevalent in pediatric patients. These include minor events (oxygen desaturation, airway obstruction, cough, or wheezing) and major events (laryngospasm and bronchospasm). Such complications may prolong hospitalization, increase healthcare costs, and cause varying degrees of physical and psychological stress in both children and their caregivers. PRAEs are documented in up to 50% of children undergoing tonsillectomy.

Certain studies in the literature have investigated preoperative premedication strategies to reduce the incidence of postoperative respiratory adverse events. However, our literature review revealed no studies evaluating the postoperative beneficial effects of the preoperative nebulized use of the agents planned in our study. Based on this gap, we designed this study with the aim of contributing new data to the current literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study
* Patients undergoing adenoidectomy or adenotonsillectomy
* Patients with ASA physical status 1-2
* Children aged 18 months to 16 years

Exclusion Criteria:

* Patients who do not agree to participate in the study
* Patients with allergy to lidocaine or 3% NaCl
* Patients with ASA physical status 3-4
* Patients whose surgery duration exceeds 1 hour

Ages: 18 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Effect of Preoperative Nebulized Lidocaine and 3% NaCl on postoperative deoxygenation | 4 hours postoperatively
  To determine which preoperative nebulized treatment (lidocaine or 3% hypertonic saline) has a beneficial effect on at least one postoperative respiratory complication-postoperative deoxygenation in pediatric patients undergoing adenoidectomy and/or adenotonsillectomy. An oxygen saturation value of ≤94% lasting for more than 2 minutes will be considered oxygen desaturation.

SECONDARY OUTCOMES:
Effect of Preoperative Nebulized Lidocaine and 3% NaCl on cough | 4 hours postoperatively
  To determine which preoperative nebulized treatment (lidocaine or 3% hypertonic saline) has a beneficial effect on at least one postoperative respiratory complication-cough in pediatric patients undergoing adenoidectomy and/or adenotonsillectomy. Postoperative cough will be assessed using a 4-point cough severity scale (0 = no cough, 1 = mild intermittent cough, 2 = frequent cough, 3 = severe or persistent cough). A score ≥2 will be considered clinically significant.
Effect of Preoperative Nebulized Lidocaine and 3% NaCl on bronkospasm | 4 hours postoperatively
  To determine which preoperative nebulized treatment (lidocaine or 3% hypertonic saline) has a beneficial effect on at least one postoperative respiratory complication-bronkospasm in pediatric patients undergoing adenoidectomy and/or adenotonsillectomy. Bronchospasm will be assessed using a 4-point bronchospasm severity scale: 0 = no bronchospasm; 1 = mild wheezing without increased respiratory effort; 2 = moderate bronchospasm with increased respiratory effort and audible wheezing; 3 = severe bronchospasm with marked respiratory distress, significant desaturation, or silent chest. A score ≥2 will be considered clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Burçin Alaçam, MD, Principal Investigator — Sakarya University

REFERENCES:
- [Background] Shen F, Zhang Q, Xu Y, Wang X, Xia J, Chen C, Liu H, Zhang Y. Effect of Intranasal Dexmedetomidine or Midazolam for Premedication on the Occurrence of Respiratory Adverse Events in Children Undergoing Tonsillectomy and Adenoidectomy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2225473. doi: 10.1001/jamanetworkopen.2022.25473. PMID 35943745
- [Background] Jarraya A, Kammoun M, Cherif O, Khcherem J, Abdelhedi A, Mhiri R. Preoperative nebulised lidocaine for children with mild symptoms of upper respiratory tract infections: A randomised controlled trial. J Perioper Pract. 2025 Jun;35(6):278-284. doi: 10.1177/17504589241276651. Epub 2024 Sep 18. PMID 40396523